CLINICAL TRIAL: NCT05676346
Title: Prevalence Study of Genetic DAO Deficiency and Lower Urinary Tract Symptoms
Brief Title: Genetic DAO Deficiency and Lower Urinary Tract Symptoms
Acronym: DAO-LUTS
Status: Completed | Type: Observational
Sponsor: Complexo Hospitalario Universitario de A Coruña (Other)
Responsible Party: Principal Investigator, José Luis Ponce Díaz-Reixa, Prinicipal Investigador. Head of Section. Urology Department., Complexo Hospitalario Universitario de A Coruña
Other Study IDs: DAO-LUTS
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Lower Urinary Tract Symptoms; Histamine Intolerance
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Oral mucosal swab Genetic single nucleotide polymorphisms rs2052129, rs10156191, rs1049742 and rs1049793
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LUTS: Patients with lower urinary tract symptoms with CACV > 3 and/or IPSS > 7.
  Interventions: Genetic: LUTS

INTERVENTIONS:
Genetic: LUTS — Patients included in this group are subjects with lower urinary tracto symptoms. An oral mucosa swab will be used to extract a genetic specimen

SUMMARY:
The aim of this study is to determinate the prevalence os genetic DAO deficiency in patients with lower urinary tract symptoms.

DETAILED DESCRIPTION:
Lower urinary tract symptoms (LUTS) encompass different symptoms and different causes, but their mechanism and etiology are not well defined. They have a high prevalence and cause discomfort and alter the quality of life. It has usually been considered that they are associated with advanced age and most scientific studies and clinical guidelines are aimed at these patients. However, many young patients show symptoms that alter their voiding quality of life. The etiology is multifactorial, the causes being attributed to bladder dysfunction and its emptying; including the prostate, urethra, and sphincter; the neurological innervation of the lower urinary tract, and medical co-morbidities. In the EPIC study, they observed that the prevalence of LUTS increases with age, from 51% in the 18-39 age group, 62% between 40-59 years, and up to 80% in patients older than 60 years. In young people, carrying disorders were more common (37.5%) than voiding symptoms (19.9%)

The etiology of the symptoms in young patients has been related to overactive bladder (OAB), benign hyperplasia (BPH), bladder neck dysfunction, urethral stenosis, drug abuse, and/or neurological disorders. Because the underlying causes are not fully known and cannot be reversed, most prevention advice is scarce. The clinical guidelines provide recommendations for lifestyle changes: fluid restriction in the hours before sleep, avoiding stimulating drinks, distraction techniques, bladder training, and pelvic floor exercises, chronic medication review and schedule readjustment, reduction weight (in case of overweight), treatment of constipation and adequate fluid intake during the day. Despite this, very few patients can improve their symptoms with these recommendations. The next step of treatment already becomes pharmacological; where alpha-blockers, anticholinergics, antimuscarinics, betamimetics, and 5 alpha-reductase inhibitors come into action. These treatments may be useful in certain patients, but in young people, failure is the norm, and surgery is often required. Both therapies imply morbidity associated with the patient, who has to deal with adverse effects, dependence on a drug for their quality of life, and the consequent economic expense. At the health level, the cost is high; It supposes a significant consumption of human, temporal, and economic resources, in progression due to the increasing prevalence and aging of the population.

The enzyme diamine oxidase (DAO) is an enzyme encoded by the AOC1 gene (OMIM#104610), located on chromosome 7 (7q-34-36). It is a secretory protein stored in vesicular structures of the plasma membrane. It is responsible for the degradation of extracellular histamine (Novotny et al., 1994, Chassande et al., 1994). In mammals, DAO is mainly expressed in the small intestine and localized to intestinal villi. Reduced histamine degradation as a consequence of low concentration or impaired activity of DAO may lead to its accumulation in plasma and the occurrence of a wide range of adverse effects due to the ubiquitous distribution of histamine receptors in different organs and tissues.

It is estimated that DAO deficiency affects 15% of the general population, according to clinical practice. It may have a genetic background. In this sense, the polymorphisms of the gene that encodes DAO have been analyzed in-depth, and more than 50 non-synonymous single nucleotide polymorphisms (SNPs) have been identified that can alter its activity. The three most relevant SNPs affecting Caucasian individuals and leading to a reduction in their enzymatic activity are c.47C>T (rs10156191), c.995C>T (rs1049742), c.1990C>G (rs1049793). The following frequencies have been described for these AOC1 variants (95% confidence interval) among Spanish Caucasian individuals: rs10156191, 25.4% (20.16-30.58), rs1049742, 6.3% (3.42 -9.26) and rs1049793, 30.6% (25.1 -36.1).

In addition, another SNP present in the promoter region of the AOC1 gene has also been identified, with a frequency of 41.7%, which has been associated with a decrease in DAO transcriptional activity: c.-691G>T (rs2052129).

Austrian researchers recently analyzed the clinical manifestations expressed by patients diagnosed with DAO deficiency. They described a wide range of symptoms involving the gastrointestinal tract, nervous and cardiovascular systems, in addition to respiratory and dermatological symptoms. Regarding the nervous system, in patients with a confirmed diagnosis of migraine, DAO deficiency has a prevalence of 87%. At the same time, preliminary data have shown a prevalence of around 77% in a pediatric cohort of Attention Deficit Hyperactivity Disorder (ADHD) and 75% in patients with clinically diagnosed fibromyalgia. Histamine is involved in the urinary tract, affecting not only the detrusor but also the lamina propria and the urothelium. It causes an increase in muscle tension and the frequency and amplitude of spontaneous contractions. Histamine has recently also been shown to affect bladder sensation, affecting spinal sensory afferents and causing sensory urgency.

The objective of this study is to estimate the prevalence of DAO deficiency in patients with LUTS and to explore the potential role of histamine accumulation in the pathophysiology of these symptoms.

ELIGIBILITY:
Inclusion Criteria:

* CACV socre > 3 and/or
* IPSS score > 7

Exclusion Criteria:

* Pharmacological treatment for LUTS in the 2 weeks prior to study inclusion (anticholinergics, antimuscarinics, or betamimetics).
* History of previous bladder and/or prostate surgery.
* History of bladder tumor in the previous 3 months.
* History of intravesical chemotherapy in the previous 3 months.
* Active urinary tract infection in the previous 2 weeks.
* Antihistamine treatment
* History of colorectal surgery and/or previous abdomino-perineal amputation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who attend Urology outpatient clinics for lower urinary tract symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Genetic DAO deficiency prevalence | Baseline
  To estimate the prevalence of genetic diamine oxidase (DAO) deficiency in patients with lower urinary tract symptoms (LUTS).

SECONDARY OUTCOMES:
Descriptive data and genotype correlation | Baseline
  To correlate age, sex, and lower urinary tract symptoms and their severity and DAO deficiency.
Histamine intolerance and lower urinary tract symptoms correlation | Last 30 days
  Assess the coexistence of histamine intolerance symptoms and lower urinary tract symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Jose Luis Ponce Diaz-Reixa, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Undecided